CLINICAL TRIAL: NCT06165588
Title: Proteomic and Physiological Markers of Exercise-induced Physiological Stress and Fatigue in Grand Tour Cycling
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Chiel Poffé, Principal Investigator, KU Leuven
Other Study IDs: S63402
Record Dates: First submitted 2023-08-31; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Exercise Fatigue
Keywords: Cycling; Proteomics; Grand tour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cyclists: Elite cyclists participating in the Tour de France
  Interventions: Other: Tour de France

INTERVENTIONS:
Other: Tour de France — Participating in the Tour de France as cyclist

SUMMARY:
This project aims to identify the effect of a 3-week grand tour (e.g. Tour de France) on physiological markers and the blood proteome in world-class cyclists.

DETAILED DESCRIPTION:
Blood samples will be collected in world-tour cyclists in the fasted state (i) before, (ii) on the first resting day, (ii) on the second resting day, and (iv) on the final day of the Tour de France. Samples collected before and on the final day will be analyzed by proteomics, while sample from all timepoints will be assessed for specific cytokines to identify physiological markers of fatigue. In addition, questionnaires will be used to evaluate subjective feelings of fatigue and appetite.

ELIGIBILITY:
Inclusion Criteria:

* Cyclist participating in the Tour de France

Exclusion Criteria:

* Younger than 18years old

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects participating in Tour de France
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Serum proteome abundance of cyclists during Tour de France | Start of the Tour de France (day 0) - last day of the Tour de France (day 23)
  Change in serum proteome between start and end of Tour de France
Serum GDF15 (Growth and differentiation factor 15) concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Serum GDF15 throughout the grand tour
Blood haemoglobin concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Haematological profile of cyclists

SECONDARY OUTCOMES:
Serum Leptin concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Serum leptin
Red blood cell concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Red blood cells
White blood cell concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  White blood cells
Serum ghrelin concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Blood ghrelin
Serum FGF21 (fibroblast growth factor 21) concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Blood FGF21
Serum free BDNF (brain-derived neutrophic factor) concentration | Start of the Tour de France (day 0) - restday 1 (day 11) - restday 2 (day 17) - last day of the Tour de France (day 23)
  Blood BDNF

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No